CLINICAL TRIAL: NCT05568719
Title: A PHASE 3, NON-INVESTIGATIONAL PRODUCT, MULTI COUNTRY COHORT STUDY TO DESCRIBE THE LONG-TERM SAFETY AND EFFECTIVENESS OF A PRIOR SINGLE-DOSE TREATMENT WITH INVESTIGATIVE GIROCTOCOGENE FITELPARVOVEC OR FIDANACOGENE ELAPARVOVEC IN PARTICIPANTS WITH HEMOPHILIA A OR HEMOPHILIA B, RESPECTIVELY
Brief Title: Safety and Effectiveness of Giroctocogene Fitelparvovec or Fidanacogene Elaparvovec in Patients With Hemophilia A or B Respectively
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C0371017; NCT05568719 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: bleeding; adeno-associated virus based vector; gene therapy; giroctocogene fitelparvovec; fidanacogene elaparvovec; factor VIII; factor IX
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Non-investigational study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hemophilia A / giroctocogene fitelparvovec (Other): Participants have received treatment with giroctocogene fitelparvovec in a previous study and are not receiving any investigational product in this study
  Interventions: Diagnostic Test: Testing of hepatic AAV Vector integration
- Hemophilia B / fidanacogene elaparvovec (Other): Participants have received treatment with fidanacogene elaparvovec in a previous study and are not receiving any investigational product in this study
  Interventions: Diagnostic Test: Testing of hepatic AAV Vector integration

INTERVENTIONS:
Diagnostic Test: Testing of hepatic AAV Vector integration — Evaluation of AAV vector integration in participants for whom a sample of liver has been obtained through biopsy or surgical resection when clinically indicated

SUMMARY:
A study to learn about the long-term safety and efficacy of giroctocogene fitelparvovec or fidanacogene elaparvovec in patients with hemophilia A or hemophilia B respectively, who have received treatment through prior participation in a Pfizer-sponsored clinical trial. Data collection and participant visits will be based on standard of care.

ELIGIBILITY:
Inclusion Criteria:

-Only participants who received investigational giroctocogene fitelparvovec or fidanacogene eleparvovec and were enrolled in a Pfizer-sponsored study (C0371002, C0371003, C0371005, C3731001, C3731003) are eligible.

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 263 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2040-02-25 (Estimated); Study Completion 2040-02-25 (Estimated)

PRIMARY OUTCOMES:
Incidence of thromboembolic events | Day 1 to 10 years
Incidence of factor inhibitor development | Day 1 to 10 years
  FIX inhibitor development was defined as an inhibitor titer >= 0.6 Bethesda units per milliliter (BU/mL).
Incidence of hepatic malignancy | Day 1 to 10 years
Incidence of liver abnormalities | Day 1 to 10 years
Factor activity level | Day 1 to 10 years
  Factor activity level will be reported. Factor levels may be measured using different assay methods including a one-stage assay or by chromogenic substrate assay and a second one-stage assay.

SECONDARY OUTCOMES:
Total ABR (treated or untreated; (excluding bleeds related to surgery) | Day 1 to 10 years
  ABR (Annual Bleed Rate): number of bleeding episodes per year. This includes treated and untreated bleeds.
  The ABR or the annualized number of bleeding episodes per year, will be derived for each participant for each observation period by using the following formula:
  ABR = (Number of bleeds / Days in observation period) x 365.25 days/year.
Incidence of and time from vector infusion to resumption of prophylaxis | Day 1 to 10 years
  Describe incidence of resumption of prophylaxis resumption and the time (in days) to resumption of prophylaxis after receiving vector infusion.
AIR of exogenous factor (excluding infusions related to surgery) | Day 1 to 10 years
  The AIR or the annualized number of FIX infusions per year, will be derived for each participant for each observation period by using the following formula:
  AIR = (Number of FIX infusions / Days in observation period) x 365.25 days/year.
Consumption of exogenous factor (excluding infusions related to surgery) | Day 1 to 10 years
  The annualized TFC in international units (IU) will be derived for each participant for each observation period using the following formula:
  Annualized TFC = (Total units of FIX infused (IU)/ Days in observation period) x 365.25 days/year
Incidence of Non-hepatic malignancy | Day 1 to 10 years
Incidence of Auto-immune disorders | Day 1 to 10 years
Incidence of SAEs | Day 1 to 10 years
  An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly; development of a clinical thrombotic event; development of factor inhibitor; development of a hepatic malignancy; development of drug-related elevated hepatic transaminases that fail to improve with immunosuppressive regimens; occurrence of a malignancy with reasonable possibility of being related to study drug.
All cause mortality | Day 1 to 10 years
  All-cause mortality was defined as the death due to any cause during the course of study. Incidence rate was defined as the total number of participants with admissible events divided by the total (for all qualifying participants) time at risk for the cohort/treatment group of interest. Incidence rate of all-cause deaths was reported in this outcome measure.
EQ-5D-5L dimension and VAS scores | Day 1 to 10 years
  The EQ-5D-5L comprises a 5-item health status measure and a visual analog rating scale/feeling thermometer. Using the 5-dimensional Health State Classification, participants are asked to respond to five questions on different aspects of their health status that assess the following:
  1. Mobility
  2. Self-care
  3. Usual activities
  4. Pain/Discomfort
  5. Anxiety/Depression

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (10):
  - UC Davis Health, Sacramento, California
  - UC Davis Ambulatory Care Clinic, Sacramento, California
  - UC Davis Hemophilia Treatment Center, Sacramento, California
  - UC Davis Medical Center, Sacramento, California
  - UCSF Outpatient Hematology Clinic, San Francisco, California
  - USF Health Morsani Center For Advanced Healthcare, Tampa, Florida
  - Mississippi Center For Advanced Medicine, Madison, Mississippi
  - Weill Cornell Medical College-New York Presbyterian Hospital, New York, New York
  - The Childrens Hospital of Philadelphia Division of Hematology, Philadelphia, Pennsylvania
  - Washington Institute for Coagulation, Seattle, Washington
- Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia
- Ege Universitesi Hastanesi, Izmir, İ̇zmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Background] Berntorp E, Shapiro AD. Modern haemophilia care. Lancet. 2012 Apr 14;379(9824):1447-56. doi: 10.1016/S0140-6736(11)61139-2. Epub 2012 Mar 27. PMID 22456059
- [Background] WFH guidelines: https://www1.wfh.org/publication/files/pdf-1472.pdf
- [Background] Blanchette VS, Key NS, Ljung LR, Manco-Johnson MJ, van den Berg HM, Srivastava A; Subcommittee on Factor VIII, Factor IX and Rare Coagulation Disorders of the Scientific and Standardization Committee of the International Society on Thrombosis and Hemostasis. Definitions in hemophilia: communication from the SSC of the ISTH. J Thromb Haemost. 2014 Nov;12(11):1935-9. doi: 10.1111/jth.12672. Epub 2014 Sep 3. No abstract available. PMID 25059285
- [Background] Blanchette VS, McCready M, Achonu C, Abdolell M, Rivard G, Manco-Johnson MJ. A survey of factor prophylaxis in boys with haemophilia followed in North American haemophilia treatment centres. Haemophilia. 2003 May;9 Suppl 1:19-26; discussion 26. doi: 10.1046/j.1365-2516.9.s1.12.x. PMID 12709033
- [Background] Lillicrap D. Extending half-life in coagulation factors: where do we stand? Thromb Res. 2008;122 Suppl 4:S2-8. doi: 10.1016/S0049-3848(08)70027-6. PMID 18929522
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0371017